CLINICAL TRIAL: NCT04154800
Title: A First-in-Human Study to Evaluate the Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single and Multiple Doses of BMS-986209 in Healthy Participants
Brief Title: A Study to Evaluate the Safety, Tolerability, Drug Levels and Drug Effects of Single and Multiple Doses of BMS-986209 in Healthy Participants
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: Quadruple | Purpose: Treatment
Other Study IDs: CV017-003
Record Dates: First submitted 2019-11-05; First posted 2019-11-07 (Actual); Last update posted 2022-01-04 (Actual); Status verified 2021-12

CONDITIONS: Health Participants
Keywords: Healthy Participants
MeSH Terms: interventions — Itraconazole; Diltiazem

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Masking Description: Parts A,B,(Participant, Care Provider, Investigator) Part C is open-labeled and a cross- over design
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Part A:SAD (Experimental): Single Ascending Dose
  Interventions: Drug: BMS-986209
- Part B: MAD (Experimental): Multiple Ascending Dose
  Interventions: Drug: BMS-986209
- Part C: DDI (Experimental): Drug-Drug Interaction
  Interventions: Drug: BMS-986209; Drug: Itraconazole; Drug: Diltiazem
- Part A (SAD) Placebo (Experimental)
  Interventions: Other: BMS-986209 Placebo
- Part B (MAD) Placebo (Experimental)
  Interventions: Other: BMS-986209 Placebo

INTERVENTIONS:
Drug: BMS-986209 — Specified Dose on Specified Days
  Arms: Part A:SAD; Part B: MAD; Part C: DDI
Other: BMS-986209 Placebo — Specified Dose on Specified Days
  Arms: Part A (SAD) Placebo; Part B (MAD) Placebo
Drug: Itraconazole — Specified Dose on Specified Days
  Arms: Part C: DDI
Drug: Diltiazem — Specified Dose on Specified Days
  Arms: Part C: DDI

SUMMARY:
The purpose of this study is to investigate the safety and tolerability of BMS-986209 in healthy participants. The first-in-human study is designed in 3 parts that vary based on duration and food effect.

ELIGIBILITY:
For more information regarding Bristol-Myers Squibb Clinical Trial participation, please visit www.BMSStudyConnect.com.

Inclusion Criteria:

* Healthy male and female participants (not of childbearing potential) as determined by no deviation considered significant by the investigator from normal in medical history, physical examination, 12-lead ECG measurements, and clinical laboratory determinations
* Women and men must agree to follow specific methods of contraception if applicable.
* Body mass index (BMI) 18.0 to 32.0 kg/m2, inclusive. BMI = weight (kg)/(height [m])2 for participants

Exclusion Criteria:

* Women who are of childbearing potential
* Women who are breastfeeding
* Any acute or chronic medical illness
* History of dizziness and/or recurrent headaches (ie, daily headaches lasting for a 1-week duration in the last month prior to study treatment administration)
* History of heart disease or conduction disorders
* Head injury in the last 2 years, intracranial tumor, or aneurysm
* Known abdominal aneurysm
* Current or history of rectal bleeding, hematemesis, or hematuria

Other protocol-defined inclusion/exclusion criteria apply

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 114 (Actual)
Dates: Start 2019-12-06 (Actual); Primary Completion 2021-08-31 (Actual); Study Completion 2021-08-31 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events (AEs) including bleeding | Up to 18 days
Incidence of serious AEs (SAEs) | Up to 44 days
Incidence of AEs leading to discontinuation | Up to 18 days
Incidence of clinically significant changes in vital signs: Body temperature | Up to 18 days
Incidence of clinically significant changes in vital signs: Respiratory Rate | Up to 18 days
Incidence of clinically significant changes in vital signs: Seated blood pressure | Up to 18 days
Incidence of clinically significant changes in vital signs: Resting pulse rate | Up to 18 days
Incidence of clinically significant changes in electrocardiogram (ECG) parameters | Up to 18 days
Incidence of clinically significant changes in clinical laboratory tests: Hematology tests | Up to 16 days
Incidence of clinically significant changes in clinical laboratory tests: Coagulation tests | Up to 16 days
Incidence of clinically significant changes in clinical laboratory tests: Serum Chemistry tests | Up to 16 days
Incidence of clinically significant changes in clinical laboratory tests: Urinalysis tests | Up to 16 days
Incidence of clinically significant changes in clinical laboratory tests: Serology tests | Up to 16 days

SECONDARY OUTCOMES:
Maximum observed plasma concentration (Cmax) of BMS-986209 | Up to 18 days
Time of Maximum observed plasma concentration (Tmax) of BMS-986209 | Up to 18 days
Terminal plasma half-life (T-Half) of BMS-986209 | Up to 18 days
Incidence of Adverse Events (AEs) including bleeding | Up to 18 days
Incidence of serious AEs (SAEs) | Up to 44 days
Incidence of AEs leading to discontinuation | Up to 18 days
Incidence of clinically significant changes in vital signs: Body temperature | Up to 18 days
Incidence of clinically significant changes in vital signs: Respiratory Rate | Up to 18 days
Incidence of clinically significant changes in vital signs: Seated blood pressure | Up to 18 days
Incidence of clinically significant changes in vital signs: Resting pulse rate | Up to 18 days
Incidence of clinically significant changes in electrocardiogram (ECG) parameters | Up to 18 days
Incidence of clinically significant changes in clinical laboratory tests: Hematology tests | Up to 16 days
Incidence of clinically significant changes in clinical laboratory tests: Coagulation tests | Up to 16 days
Incidence of clinically significant changes in clinical laboratory tests: Serum Chemistry tests | Up to 16 days
Incidence of clinically significant changes in clinical laboratory tests: Urinalysis tests | Up to 16 days
Incidence of clinically significant changes in clinical laboratory tests: Serology tests | Up to 16 days
Percent change from baseline in plasma activated partial thromboplastin time (aPTT) levels | Up to 16 days
Percent change from baseline in factor XI (FXI) clotting activity | Up to 16 days

CONTACTS AND LOCATIONS:
Overall Officials: Bristol-Myers Squibb, Study Director — Bristol-Myers Squibb
Locations (1):
- PPD Development, LP, Austin, Texas, United States

REFERENCES:
- See also: BMS Clinical Trial Information — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: BMS Clinical Trial Patient Recruiting — https://www.bmsstudyconnect.com/s/US/English/USenHome
- See also: Investigator Inquiry Form — https://www.bms.com/researchers-and-partners/clinical-trials-and-research.html
- See also: FDA Safety Alerts and Recalls — https://www.fda.gov/Safety/MedWatch/SafetyInformation/default.htm